CLINICAL TRIAL: NCT03430362
Title: Effect Of Intravenous Hyoscine -N-Butyl Bromide In Management Of Prolonged Labor In Nulliparous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Prolonged Labor
MeSH Terms: interventions — Butylscopolammonium Bromide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Group A will receive injection Hyoscine butyl bromide 20 mg first dose at the time of amniotomy, and second dose 2 hours after. Group B, will receive normal saline same volume first dose at the time of amniotomy, and second dose 2 hours after
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyoscine group (Active Comparator): 7. Group A will receive injection Hyoscine butyl bromide 40 mg single intravenous dose
  Interventions: Drug: Hyoscine N Butylbromide
- Control group (Placebo Comparator): Group B, will receive 2 ml of normal saline single intravenous dose
  Interventions: Drug: Normal Saline 0.9%

INTERVENTIONS:
Drug: Hyoscine N Butylbromide — 7. Group A will receive injection Hyoscine butyl bromide 40 mg single intravenous dose
  Other Names: Buscopan
  Arms: Hyoscine group
Drug: Normal Saline 0.9% — Group B, will receive 2 ml of normal saline single intravenous dose
  Other Names: Saline
  Arms: Control group

SUMMARY:
Women will be admitted when active phase of labour starts defined as the presence of at least three regular uterine contractions over 10 minutes with cervical dilatation four centimeters with cervical effacement not less than 50% and no progress of labor for 2 hours or more.

Amniotomy was done in those with intact membrane and continuous electronic fetal monitoring was done. Women with prolonged labor after these measures were randomly divided using automated web-based randomization system into 2 equal groups. Group I included 50 women received 40mg HBB (Buscopan, Memphis Co, Giza, Egypt) intravenous bolus injection. Group II included 50 women received 2 ml of normal saline. The obstetrician, participants and outcome assessor were all blinded to the group assignment. Labor will be monitored by Vaginal examination every two hours. The duration of the first stage was calculated from the time of cervical dilatation of three to four centimeters in active labor until a fully dilated cervix was observed.

DETAILED DESCRIPTION:
Women will be admitted when active phase of labour starts defined as the presence of at least three regular uterine contractions over 10 minutes with cervical dilatation four centimeters with cervical effacement not less than 50% and no progress of labor for 2 hours or more.

Amniotomy was done in those with intact membrane and continuous electronic fetal monitoring was done. Women with prolonged labor after these measures were randomly divided using automated web-based randomization system into 2 equal groups. Group I included 50 women received 40mg HBB (Buscopan, Memphis Co, Giza, Egypt) intravenous bolus injection. Group II included 50 women received 2 ml of normal saline. The obstetrician, participants and outcome assessor were all blinded to the group assignment. Labor will be monitored by Vaginal examination every two hours. The duration of the first stage was calculated from the time of cervical dilatation of three to four centimeters in active labor until a fully dilated cervix was observed.

ELIGIBILITY:
Inclusion Criteria:

* • Nulliparous women.

  * cervical dilatation in the active phase of less than 1.2 cm/h for nulliparous women
  * Gestational age ≥ 37 weeks.
  * Singleton pregnancy.
  * Vertex presentation.
  * Cervical dilatation ≥ 4cm.
  * No evidence of maternal or fetal distress.
  * Average size baby.

Exclusion Criteria:

* History of cervical surgery.
* Mal-presentation and mal-positions.
* Hypersensitivity to Hyoscine.
* Contraindication for vaginal delivery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-02-16 (Actual)

PRIMARY OUTCOMES:
the duration of active phase of first stage of labor | 8 hours after hyoscine adminstration
  time elapsed between start of active phase till full cervical dilatation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Sorour EH, ElSadek MM, Hassan SM, Shoab AY. A randomized controlled study of the effect of hyoscine butylbromide on duration of labor in primigravida women with prolonged labor. Arch Gynecol Obstet. 2021 Dec;304(6):1513-1518. doi: 10.1007/s00404-021-06087-7. Epub 2021 May 13. PMID 33983512